CLINICAL TRIAL: NCT05855785
Title: Effect of Dual-task Exercise on Cognitive and Physical Function in the Elderly With Mild Cognitive Impairment: a Randomized Controlled Trial
Brief Title: Effect of Dual Task Exercise on Cognitive and Physical Function in the Elderly With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Boramae Hospital (Other)
Collaborators: National Rehabilitation Center, Ministry of Health and Welfare, Korea (Unknown)
Responsible Party: Principal Investigator, Cha Hee Young, Principal Investigator, Seoul National University Boramae Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-2020-38
Record Dates: First submitted 2023-03-30; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Dysfunction; Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The exercise group (Experimental): The exercise group underwent 8-week, 3 times a week, 60-minute group exercise sessions, which were comprised of moderate-to-high intensity exercise and simultaneous cognitive tasks. The exercise group also performed moderate-intensity home aerobic exercises for at least 60 minutes per week.
  Interventions: Behavioral: dual task exercise
- The control group (Other): The control group performed 60-minute light intensity home exercise, 4 times a week for 8 weeks.
  Interventions: Behavioral: home exercise

INTERVENTIONS:
Behavioral: dual task exercise — 8-week, 3 times a week, 60-minute group exercise sessions, which were comprised of moderate-to-high intensity exercise and simultaneous cognitive tasks
  Arms: The exercise group
Behavioral: home exercise — 60-minute light intensity home exercise, 4 times a week for 8 weeks
  Arms: The control group

SUMMARY:
The purpose of this study is to investigate the effect of the dual task exercise program on cognitive and physical function in the elderly with mild cognitive impairment.

DETAILED DESCRIPTION:
All participants provided written informed consent before study participation. A total of 12 community-dwelling participants were randomized either to the exercise group or to the control group.

The exercise group underwent 8-week, 3 times a week, 60-minute group exercise sessions, which were comprised of moderate-to-high intensity exercise and simultaneous cognitive tasks. They also performed moderate-intensity home aerobic exercises for at least 60 minutes per week. The control group performed 60-minute light intensity home exercise, 4 times a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* a score on the Korean Montreal Cognitive Assessment (MoCA-K) of 25 points or below
* aged 65 or more
* no physical or medical problem which impairs moderate to vigorous physical activity

Exclusion Criteria:

* uncontrolled or unstable cardiovascular disease
* malignancy affecting general condition
* musculoskeletal problems affecting motor performance
* speech and hearing impairment
* other organic brain diseases

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-04-08 (Actual)

PRIMARY OUTCOMES:
Dual task cost in Timed up and go (TUG) | Baseline
  Participants completed both single-task (ST) and dual-task (DT) tests at baseline and post-intervention.
  For a ST condition, participants performed motor task only such as Timed up and go (TUG). TUG measured the time of taking to rise from a chair, walking three meters, turning around 180 degrees, walking back to the chair, and sitting down while turning 180 degrees. For a DT condition, participants performed TUG while performing serial 3 simultaneously. Serial 3 is descending subtraction task, where the patient counts down from one hundred by threes. In the DT condition, participants were given no instruction regarding the prioritization of one task over the other. We calculated TUG duration in both conditions. Dual task cost(DTC) were calculated as a percentage as follows: (%DTC) = [dual task duration or speed - single task duration or speed] / [single task duration or speed] * 100%. The lower DTC indicates efficiency in cognitive-motor interplay and good dual task ability.
Dual task cost in 10-meter walking test | Baseline
  Participants completed both single-task (ST) and dual-task (DT) tests at baseline and post-intervention.
  For a ST condition, participants performed motor task only such as 10-meter walking test (10MWT). 10MWT is a performance measure used to assess walking speed over a short distance. For a DT condition, participants performed 10MWT while performing serial 3 simultaneously. Serial 3 is descending subtraction task, where the patient counts down from one hundred by threes. In the DT condition, participants were given no instruction regarding the prioritization of one task over the other. We calculated 10MWT gait speed in both conditions. Dual task cost(DTC) were calculated as a percentage as follows: (%DTC) = [dual task duration or speed - single task duration or speed] / [single task duration or speed] * 100%. The lower DTC indicates efficiency in cognitive-motor interplay and good dual task ability.
Dual task cost in Timed up and go (TUG) | immediately after the 8-week intervention
  Participants completed both single-task (ST) and dual-task (DT) tests at baseline and post-intervention.
  For a ST condition, participants performed motor task only such as Timed up and go (TUG). TUG measured the time of taking to rise from a chair, walking three meters, turning around 180 degrees, walking back to the chair, and sitting down while turning 180 degrees. For a DT condition, participants performed TUG while performing serial 3 simultaneously. Serial 3 is descending subtraction task, where the patient counts down from one hundred by threes. In the DT condition, participants were given no instruction regarding the prioritization of one task over the other. We calculated TUG duration in both conditions. Dual task cost(DTC) were calculated as a percentage as follows: (%DTC) = [dual task duration or speed - single task duration or speed] / [single task duration or speed] * 100%. The lower DTC indicates efficiency in cognitive-motor interplay and good dual task ability.
Dual task cost in 10-meter walking test | immediately after the 8-week intervention
  Participants completed both single-task (ST) and dual-task (DT) tests at baseline and post-intervention.
  For a ST condition, participants performed motor task only such as 10-meter walking test (10MWT). 10MWT is a performance measure used to assess walking speed over a short distance. For a DT condition, participants performed 10MWT while performing serial 3 simultaneously. Serial 3 is descending subtraction task, where the patient counts down from one hundred by threes. In the DT condition, participants were given no instruction regarding the prioritization of one task over the other. We calculated 10MWT gait speed in both conditions. Dual task cost(DTC) were calculated as a percentage as follows: (%DTC) = [dual task duration or speed - single task duration or speed] / [single task duration or speed] * 100%. The lower DTC indicates efficiency in cognitive-motor interplay and good dual task ability.

SECONDARY OUTCOMES:
Korean Montreal Cognitive Assessment (MoCA-K) | Baseline
  MoCA-K is a screening test to assess cognitive functions such as attention, concentration, execution, memory, vocabulary, visual space, abstraction, and calculation. MoCA-K is a test for mild cognitive impairment and it takes about 10 minutes to run. It assesses cognitive functions such as attention, concentration, execution, memory, vocabulary, visual space, abstraction, calculation and support. Of a maximum 30 points, a score of 25 or higher is considered normal.
Korean Montreal Cognitive Assessment (MoCA-K) | immediately after the 8-week intervention
  MoCA-K is a screening test to assess cognitive functions such as attention, concentration, execution, memory, vocabulary, visual space, abstraction, and calculation. MoCA-K is a test for mild cognitive impairment and it takes about 10 minutes to run. It assesses cognitive functions such as attention, concentration, execution, memory, vocabulary, visual space, abstraction, calculation and support. Of a maximum 30 points, a score of 25 or higher is considered normal.
Korean Mini Mental Status Examination (K-MMSE) | Baseline
  K-MMSE is a screening test for dementia that can evaluate various areas of cognitive function in a short time of 5 to 10 minutes such as time orientation, place orientation, memory, attention and calculation, understanding and judgment, and language. Of a maximum 30 points, a score of less than 24 is considered dementia.
Korean Mini Mental Status Examination (K-MMSE) | immediately after the 8-week intervention
  K-MMSE is a screening test for dementia that can evaluate various areas of cognitive function in a short time of 5 to 10 minutes such as time orientation, place orientation, memory, attention and calculation, understanding and judgment, and language. Of a maximum 30 points, a score of less than 24 is considered dementia.
Computerized cognitive test(digit span test, visual learning test, verbal learning test, the Stroop Color and Word test, Boston naming test, trail making test, and verbal fluency test) | Baseline
  Computerized cognitive test is a test method which quantitatively measures patients' cognitive problems in a systematic and standardized manner using a computer. Various neurocognitive function tests such as attention, memory, memory-motor coordination, and comprehensive cognitive thinking ability are possible through computerized cognitive test. Card sorting test, digit span test, visual learning test, verbal learning test, and Stroop word color test were conducted for precise cognitive function evaluation.
Computerized cognitive test(digit span test, visual learning test, verbal learning test, the Stroop Color and Word test, Boston naming test, trail making test, and verbal fluency test) | immediately after the 8-week intervention
  Computerized cognitive test is a test method which quantitatively measures patients' cognitive problems in a systematic and standardized manner using a computer. Various neurocognitive function tests such as attention, memory, memory-motor coordination, and comprehensive cognitive thinking ability are possible through computerized cognitive test. Card sorting test, digit span test, visual learning test, verbal learning test, and Stroop word color test were conducted for precise cognitive function evaluation.
Short Physical Performance Battery (SPPB) | Baseline
  SPPB is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people . The scores range from 0 (worst performance) to 12 (best performance).
Short Physical Performance Battery (SPPB) | immediately after the 8-week intervention
  SPPB is a group of measures that combines the results of the gait speed, chair stand and balance tests. It has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people . The scores range from 0 (worst performance) to 12 (best performance).
Berg Balance Scale (BBS) | Baseline
  BBS is an evaluation tool designed to measure the balance of the elderly and consists of 56 points in 14 items that apply daily life movements. It is a measure to objectively evaluate static and dynamic balance ability in various postures such as sitting, standing, and posture change. Higher score means well balance function.
Berg Balance Scale (BBS) | immediately after the 8-week intervention
  BBS is an evaluation tool designed to measure the balance of the elderly and consists of 56 points in 14 items that apply daily life movements. It is a measure to objectively evaluate static and dynamic balance ability in various postures such as sitting, standing, and posture change. Higher score means well balance function.
Falls Efficacy Scale (FES) | Baseline
  FES is a questionnaire that evaluates the confidence to perform the activities without falling from the 10 activities. Higher score means good function.
Falls Efficacy Scale (FES) | immediately after the 8-week intervention
  FES is a questionnaire that evaluates the confidence to perform the activities without falling from the 10 activities. Higher score means good function.
Activities-specific Balance Confidence (ABC) | Baseline
  ABC consists of 16 surveys and it evaluates level of self-confidence in doing the activity without losing balance or becoming unsteady by choosing one of the percentage points on the scale from 0% to 100%.
Activities-specific Balance Confidence (ABC) | immediately after the 8-week intervention
  ABC consists of 16 surveys and it evaluates level of self-confidence in doing the activity without losing balance or becoming unsteady by choosing one of the percentage points on the scale from 0% to 100%.
Grip strength | Baseline
  Grip strength was measured by hand dynamometer for evaluating muscle strength. It is measured using pound(lb).
Grip strength | immediately after the 8-week intervention
  Grip strength was measured by hand dynamometer for evaluating muscle strength. It is measured using pound(lb).
Korean version of Physical Activity Scale for the Elderly (K-PASE) | Baseline
  K-PASE measures various physical activities of the elderly which are divided into sedentary life, leisure time activities, housework activities, and work-related activities. The score is calculated by multiplying the level and frequency of each activity using the conversion table. Higher score means higher activity.
Korean version of Physical Activity Scale for the Elderly (K-PASE) | during intervention(8 weeks)
  K-PASE measures various physical activities of the elderly which are divided into sedentary life, leisure time activities, housework activities, and work-related activities. The score is calculated by multiplying the level and frequency of each activity using the conversion table. Higher score means higher activity.
International Physical Activity Questionnaires Short form (IPAQ) | Baseline
  IPAQ Short form consists of 7 surveys and evaluate the degree of physical activity and the time spent on physical activity for one week.
International Physical Activity Questionnaires Short form (IPAQ) | during intervention (8 weeks)
  IPAQ Short form consists of 7 surveys and evaluate the degree of physical activity and the time spent on physical activity for one week.
Metabolic Equivalent Task (MET) minutes per week | Baseline
  MET minutes per week were evaluated to measure the degree of physical activity before intervention and every week during 8 weeks of intervention. MET minutes per week was calculated based on IPAQ.
Metabolic Equivalent Task (MET) minutes per week | during intervention(8 weeks)
  MET minutes per week were evaluated to measure the degree of physical activity before intervention and every week during 8 weeks of intervention. MET minutes per week was calculated based on IPAQ.
Bioelectrical Impedance Analysis | Baseline
  Bioelectrical Impedance Analysis was evaluated using Inbody for changes in body composition before and after intervention. Specifically, body weight, body fat percent, body mass index (BMI), skeletal muscle mass, lean mass, fat mass, waist hip ratio were evaluated.
Bioelectrical Impedance Analysis | immediately after the 8-week intervention
  Bioelectrical Impedance Analysis was evaluated using Inbody for changes in body composition before and after intervention. Specifically, body weight, body fat percent, body mass index (BMI), skeletal muscle mass, lean mass, fat mass, waist hip ratio were evaluated.
Exercise Identity Scale (EIS) | Baseline
  Exercise Identity Scale (EIS) is a measure of how important exercise is in daily life
Exercise Identity Scale (EIS) | immediately after the 8-week intervention
  Exercise Identity Scale (EIS) is a measure of how important exercise is in daily life
Psychological Need Satisfaction in Exercise Scale (PNSE) | Baseline
  Psychological Need Satisfaction in Exercise Scale (PNSE) is an exercise psychological measure consisting of detailed items of self-confidence, autonomy, and belonging related to exercise.
Psychological Need Satisfaction in Exercise Scale (PNSE) | immediately after the 8-week intervention
  Psychological Need Satisfaction in Exercise Scale (PNSE) is an exercise psychological measure consisting of detailed items of self-confidence, autonomy, and belonging related to exercise.
Godin Leisure Time Exercise Questionnaire (GLTEQ) | Baseline
  Godin Leisure Time Exercise Questionnaire (GLTEQ) is a self-report measure of the frequency of light-intensity, moderate-intensity, and vigorous-intensity leisure-time physical activity. It evaluated how satisfied the participants were with the intervention.
Godin Leisure Time Exercise Questionnaire (GLTEQ) | immediately after the 8-week intervention
  Godin Leisure Time Exercise Questionnaire (GLTEQ) is a self-report measure of the frequency of light-intensity, moderate-intensity, and vigorous-intensity leisure-time physical activity. It evaluated how satisfied the participants were with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Se Hee Jung, MD, PhD, Study Chair — Department of Rehabilitation Medicine, Seoul National University Boramae Medical Center
Locations (1):
- Seoul National University Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Plummer P, Eskes G. Measuring treatment effects on dual-task performance: a framework for research and clinical practice. Front Hum Neurosci. 2015 Apr 28;9:225. doi: 10.3389/fnhum.2015.00225. eCollection 2015. PMID 25972801